CLINICAL TRIAL: NCT02279082
Title: DFN-02 Open Label Safety Study in Patients With Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFN-02-CD-010
Record Dates: First submitted 2014-10-23; First posted 2014-10-30 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Acute Migraine
MeSH Terms: interventions — DFN-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DFN-02 (Experimental): DFN-02 to be taken during migraine attack
  Interventions: Drug: DFN-02

INTERVENTIONS:
Drug: DFN-02 — Active Experimental Drug

SUMMARY:
A multi-center, open-label, safety study of DFN-02 for the Treatment of Acute Migraines

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of acute migraine (using International Classification of Headache Disorders [ICHD] criteria, second edition);
2. Patients who, in the opinion of the investigator, are willing and able to:

   * Return to the study site within 72 hours of the first use of study medication,
   * Record each migraine and each instance of the use of study medication and rescue medication in a patient diary for the duration of the study;
3. Patients who can use the nasal spray device correctly after instruction.

Exclusion Criteria:

1. Patients on onabotulinumtoxinA (Botox®) or other botulinum toxin treatment; or history of receiving such treatment 180 days prior to screening;
2. Patients with a history of stroke or transient ischemic attack (TIA);
3. Patients with a history of migralepsy or a concurrent diagnosis of seizure disorder;
4. Patients who cannot differentiate between a migraine headache and a tension-type or cluster headache;
5. Patients with ischemic coronary artery disease (CAD; ie, angina pectoris, history of myocardial infarction or documented silent ischemia or coronary artery vasospasm, including Prinzmetal's angina);
6. Patients with Wolff-Parkinson-White syndrome or arrhythmias associated with other cardiac accessory conduction pathway disorders;
7. Patients with uncontrolled hypertension (screening systolic/diastolic blood pressure > 140/90 mmHg);
8. Patients with peripheral vascular disease or ischemic bowel disease;
9. Patients taking any medications or with illnesses likely to affect the physiology of the nasal mucosa (ie, patients with nasal septum surgery, chronic sinusitis, or chronic nasal rhinitis). (Note: Patients who have acute conditions such as acute sinusitis may be rescreened 14 days after resolution of acute sinusitis.);
10. Patients with any abnormal nasal physiology or pathology which, in the opinion of the investigator, would not allow the objectives of the study to be accomplished;
11. Patients with known intolerance to nasal sprays;
12. Patients with severe renal impairment (defined as serum creatinine > 2 mg/dL);
13. Patients with serum total bilirubin > 2.0 mg/dL;
14. Patients with serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.5 times the upper limit of normal (ULN);
15. Patients with a history of alcohol or substance abuse (including marijuana and medical marijuana) within 1 year that would compromise data collection;
16. Patients with a positive urine drug screen for illicit drugs or for prescription drugs not explained by stated concomitant medications. (Positive drug screen for marijuana is exclusionary.):

    1. Patients consuming opioids for the treatment of migraine or using opioids or barbiturates temporarily for a legitimate medical cause may participate as long as they do not meet the MOH criteria.
    2. Benzodiazepines are allowed if used for legitimate medical use.
    3. Chronic use of amphetamines to treat attention deficit disorder (ADD) or attention deficit hyperactivity disorder (ADHD) and related disorders is allowed as long as the regimen has been stable for at least 3 months prior to screening and is expected to remain stable throughout the study.

    Note: For the above-mentioned conditions, the site must obtain medical monitor approval.
17. Patients with a history of or current neurological or psychiatric impairment, or cognitive dysfunction that, in the opinion of the investigator, would compromise data collection;
18. Patients who have received treatment with an investigational drug or device within 4 weeks of the screening visit or participated in a central nervous system clinical trial in the 3 months prior to screening;
19. Patients who test positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody serology testing.
20. Patients with any other medical condition that, in the judgment of the investigator or medical monitor, would confound the objectives of the study (eg, cancer history [except basal cell carcinoma], systemic lupus erythematosus)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Arizona Research Center, Phoenix, Arizona
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Northern California Clinical Research Center, Redding, California
  - Breakthrough Clinical Trials, San Bernardino, California
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - Florida Clinical Research Center, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Neurology Clinical Research, Inc, Sunrise, Florida
  - Carman Research, Smyrna, Georgia
  - Novex Clinical Research, New Bedford, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurologic Institute, Amherst, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - Community Research, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - FutureSearch Trials of Neurology, LP, Austin, Texas
  - Protenium Clinical Research, LLC, Bedford, Texas
  - Future Search Trials of Dallas, LP, Dallas, Texas

REFERENCES:
- [Background] Munjal S, Gautam A, Offman E, Brand-Schieber E, Allenby K, Fisher DM. A Randomized Trial Comparing the Pharmacokinetics, Safety, and Tolerability of DFN-02, an Intranasal Sumatriptan Spray Containing a Permeation Enhancer, With Intranasal and Subcutaneous Sumatriptan in Healthy Adults. Headache. 2016 Oct;56(9):1455-1465. doi: 10.1111/head.12905. Epub 2016 Sep 10. PMID 27613076
- [Result] Munjal S, Brand-Schieber E, Allenby K, Spierings ELH, Cady RK, Rapoport AM. A multicenter, open-label, long-term safety and tolerability study of DFN-02, an intranasal spray of sumatriptan 10 mg plus permeation enhancer DDM, for the acute treatment of episodic migraine. J Headache Pain. 2017 Dec;18(1):31. doi: 10.1186/s10194-017-0740-3. Epub 2017 Mar 1. PMID 28251391

RESULTS

PARTICIPANT FLOW:
Groups:
- DFN-02: Active DFN-02 (Nasal Sumatriptan 10mg)
  DFN-02: Active Experimental Drug
Period: Overall Study
Arm/Group | DFN-02
Started | 167 (Intentions were to have 173 participants, but only 167 participants received study drug.)
Completed | 134
Not Completed | 33

BASELINE CHARACTERISTICS:
Groups:
- DFN-02 (Single Arm, Open Label): Active DFN-02
  DFN-02: Active Experimental Drug
Arm/Group | DFN-02 (Single Arm, Open Label)
Number analyzed (Participants) | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 167
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 25
  White | 136
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- DFN-02: Active DFN-02
  DFN-02: Active Experimental Drug
Arm/Group | DFN-02
Number analyzed (Participants) | 167
Participants | 120

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | DFN-02 (Single Arm, Open Label)
All-Cause Mortality (participants affected / at risk) | 0/167
Serious Adverse Events (participants affected / at risk) | 4/167
Other Adverse Events (participants affected / at risk) | 120/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DFN-02 (Single Arm, Open Label) (N=167)
Diverticulitis (Gastrointestinal disorders) | 1
cholecystitis (Gastrointestinal disorders) | 1
menometrorrhagia (Reproductive system and breast disorders) | 1
pyelonephritis (Renal and urinary disorders) | 1
myocardial infarction (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFN-02 (Single Arm, Open Label) (N=167)
dysgeusia (Nervous system disorders) | 35 (232)
Application site pain (General disorders) | 51 (568)
Application Site Reaction (General disorders) | 9 (32)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (24)
Nasopharyngitis (Infections and infestations) | 12 (13)
Sinusitis (Infections and infestations) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less